CLINICAL TRIAL: NCT04289974
Title: An Open, Multicenter Study for the Predicted Biomarkers of CDK4/6 Inhibitors (Palbociclib) in ER-positive Metastasis Breast Cancer
Brief Title: Predicted Biomarkers of CDK4/6 Inhibitors (Palbociclib) in ER-positive Metastasis Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: OrigiMed (Industry)
Responsible Party: Principal Investigator, Li Qiao, Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: LQ005
Record Dates: First submitted 2019-07-31; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: Palbociclib; endocrinotherapy; resistance
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Fulvestrant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Formalin fixed paraffin-embedded (FFPE) tumor tissue for DNA sequencing obtained from surgical/needle biopsy; fresh or liquid nitrogen frozen tissues for RNA sequencing obtained from surgical biopsy; peripheral blood (PB) samples for ctDNA sequencing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Palbociclib+fulvestrant: 100 cases of patients with ER+, HER2- breast cancer, experienced resistance after first line endocrinotherapy, will be assigned participants into treatment regimen, including palbociclib combined with fulvestrant.
  FFPE blocks/sections or fresh tumor tissues/biopsies will be obtained from the hospitals on the points before administration and since resistance appearance. The tissue will be sequenced by a pan-cancer DNA panel (500+ genes) and whole transcriptome sequencing (WTS).
  5-10 ml peripheral blood will be collected from each patient on the points before administration, 1 month after treatment, every subsequent visit and resistance appearance. The liquid biopsy will be sequenced by a pan-cancer ctDNA panel (300+ genes).
  The genomic characteristics of patients received resistance will be analyzed. The relevant pathway mechanisms will be identified.
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — Palbociclib (125 mg PO qDay for Days 1-21 of each 28-day cycle) combined with Fulvestrant (500 mg IM on Days 1, 15, and 29, and then once monthly thereafter)
  Other Names: Fulvestrant

SUMMARY:
This is a multi-center, observational study designed to explore the regulatory mechanism of palbociclib correlative pathways in therapeutic process of breast cancer, employing next generation sequencing (NGS) on DNA and RNA. This study also monitor the clonal evolution of genes by tracing the ctDNA.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-70 years old at the time of sign informed consent
* patients diagnosed as breast cancer with evidence supporting metastatic disease, unsuitable for radical operation or radiotherapy, with no chemotherapy indication
* full histological or cytological assessment of ER+, HER2- breast cancer
* refractory to the most recent endocrine therapy, or progression within 12 months of endocrine therapy
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1, no refractory within recent 2 weeks
* patients with at least 1 measuralbe lesion; lesions will be excluded if received radiotherapy, unless had confirmed progression
* life expectancy of 12 weeks or more
* clinical laboratory test indicators meet the following criteria:
* PLT≥100×10^9/L
* ANC≥1.5×10^9/L
* Hgb≥90 g/L
* TBil≤1.5 ULN
* ALT and AST ≤3 ULN
* creatinine≤1.5 ULN or creatinine clearance rate≥50 mL/min
* patients who signed informed consents before any projects, sampling and analysis; be available of tumor tissue biopsy and liquid biopsy; be cooperative for observation period
* patients can swallow oral drugs
* In addition to alopecia and stable peripheral neurotoxicity below grade 2, any clinical toxicity associated with previous treatment prior to enrollment must be restored to baseline or grade 1.

Exclusion Criteria:

* no prior treatment
* receiving treatment other than the trial 4 weeks prior to the study, or participating in another clinical study
* unwilling to provide tissue and blood for genetic testing
* non-resistant on endocrine therapy before treating with palbociclib
* progress of ≥ 2nd line endocrine therapy
* patients with advanced disease, symptoms, visceral spread, and life-threatening complications in the short term (including large uncontrollable spills [thoracic, pericardium, abdominal cavity], pulmonary lymphangitis, and liver involvement>50%)
* patients with active, uncontrolled or symptomatic central nervous system metastases, cancerous meningitis or clinical signs suggesting pia mater disease, brain edema and/or tumor growth. Patients with a history of central nervous system metastasis or spinal cord compression, if they have received local treatment (such as radiation therapy, stereotactic surgery) and are clinically stable, they need to stop convulsions and steroids for at least 4 weeks before randomization.
* patients received major surgery, chemotherapy, radiation therapy, or other anticancer treatments within 2 weeks prior to enrollment
* diagnosis of any other malignant tumor, within 3 years prior to the enrollment, except adequately treated basal/squamous cell skin cancer or cervical carcinoma
* assessed as not eligible to participate in the trial
* infused whole blood without leukocytes removing within 120 days prior to sampling
* during lactation or with positive blood or urine pregnancy test

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: metastatic breast cancer patients of ER+/HER2- with resistance of first line endocrine therapy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Pathway regulatory mechanism during palbociclib treatment on ER+/HER2- breast cancer. | 2 year
  Crosstalk patterns of genetic change processes with significant correlation with treatment of palbociclib combined endocrinotherapy, assessed by DNA and RNA sequencing.
Patterns of clonal changing on lesions during treatment of palbociclib combined endocrinotherapy. | 2 year
  The evolution patterns of genetic profiles since the begining of palbociclib combined endocrinotherapy until occurance of drug resistance obtained by collecting ctDNA variations dynamically.

SECONDARY OUTCOMES:
Genetic indicators of effect and prognosis of palbociclib combined endocrinotherapy on ER+/HER2- breast cancer. | 2 year
  Indicator genes with measurable up/down regulated activities of ER+/HER2- breast cancer patients significantly correlated with treatment of palbociclib combined endocrinotherapy.
Genetic indicators of resistance of palbociclib combined endocrinotherapy on ER+/HER2- breast cancer. | 2 year
  Specific genetic aberrations in alternative pathways, i.e. CCND1 amplification or RB1 inactivation, before treatment of palbociclib combining with endocrinotherapy and after drug-resistance of the breast cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, PHD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, ChineseAMS, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided